CLINICAL TRIAL: NCT01897857
Title: Influence of DM on Artery Blood Flow and Complications After Radial Artery Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2013-0209
Record Dates: First submitted 2013-07-01; First posted 2013-07-12 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Renal Disease
Keywords: diabetes mellitus(DM); radial artery cannulation; artery blood flow; complication; End stage renal disease undergoing kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic; Diabetes Mellitus | interventions — Ultrasonography, Doppler, Duplex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DM kidney transplantation (Experimental): patient with DM undergoing undergoing kidney transplantation
  Interventions: Device: duplex Doppler ultrasonography
- without DM undergoing kidney transplantation (Active Comparator): patient without DM undergoing undergoing kidney transplantation
  Interventions: Device: duplex Doppler ultrasonography

INTERVENTIONS:
Device: duplex Doppler ultrasonography

SUMMARY:
In atherosclerotic patients undergoing kidney transplantation, arterial cannulation is commonly performed for continuous monitoring of systemic blood pressure and intermittent assessment of arterial blood gases. The radial artery is the preferred artery, because of its well-documented low complication rate and easy access, but, radial artery cannulation is may associated with complications. Atherosclerosis is a systemic phenomenon, and structural changes attributable to atherosclerosis, such as luminal narrowing, intimal hyperplasia, and reduction in distensibility occur frequently throughout the arterial tree. Especially in patients with diabetes mellitus (DM), the radial artery is prone to atherosclerosis and perhaps calcification. In a recent study, it was found that the radial artery flow was decreased immediately after cannulation, but recovered to its pre-cannulation value after 5min, whereas a compensatory increase of blood flow in the ulnar artery occured immediately after cannulation, persisting until 5 min. This study enrolled the patients of ASA physical status 1-2. In the patients scheduled for elective kidney transplantation, this compensatory increase of blood flow in the ulnar artery may not be occurred, because of atherosclerosis, particularly in patients with DM. In our study, we found whether there is appropriate compensatory increase of blood flow in the ulnar artery after the radial artery cannulation in two groups, patients with DM (group DM) or without DM (group nonDM), both undergoing elective kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* age > 20yrs undergoing kidney transplantation
* ASA physical status ≥ 3
* patients with DM (DM group), patients without DM (nonDM group)

Exclusion Criteria:

* coagulopathy
* inflammation or infection at the puncture site for cannulation
* a positive result on the modified Allen's test
* the cannulation failed twice
* Acute renal allograft rejection

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
the compensatory changes in ulnar artery blood flow after radial artery cannulation | Change from Baseline in ulnar artery blood before anesthesia, before cannulation, 5 min after cannultion, 20 min after removal of the arterial catheter, 24 hous after cannulation
  to evaluate the compensatory changes in ulnar artery blood flow after radial artery cannulation using duplex Doppler ultrasonography at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, Seoul, South Korea